CLINICAL TRIAL: NCT07278401
Title: Community Pharmacies as Social Determinant of Health Navigators
Acronym: SDoH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: CPESN-NY Pharmacies (Unknown); Tops Pharmacies (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, David Matthew Jacobs, Associate Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 8733; UM1TR005296 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Social Needs Status
Keywords: Social Determinants of Health; Community Pharmacies
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: This is a single intervention group with a matched control group with a local health information exchange.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social needs screenings control group (No Intervention): Individuals within the same healthcare system that are matched based on similar characteristics.
- Social needs screenings and referrals participants (Other): Patients who have been identified to have needs via the screening survey who are referred to a community based organization by the pharmacist navigator.
  Interventions: Other: Social needs screenings and referrals

INTERVENTIONS:
Other: Social needs screenings and referrals — Community pharmacies will distribute social needs screening surveys to patients and refer them to local community based organizations based off of identified needs.
  Arms: Social needs screenings and referrals participants

SUMMARY:
Type 1 hybrid effectiveness-implementation study using a quasi-experimental, difference-in-difference (DID) design to deliver a comprehensive social needs screening and navigation program by integrating Community Health Workers (CHWs) into community pharmacies across under-resourced areas in Western New York (WNY).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 18 years
* English speaking
* Presenting to one of the participating pharmacies. For the pharmacies to be included, they must be enrolled within the Community Pharmacy Enhanced Services Network - NY (CPESN-NY) or associated with Tops Pharmacies. The pharmacies must have the ability to collaborate with Healthelink and referring partners (e.g., Wellconnected) and the staffing capacity to have a SDoH screening program with Community Health Worker Training. The pharmacies' physical address must be located within Erie County

Exclusion Criteria:

* Subjects ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Outcomes | 12 months
  Primary effectiveness outcomes in composite healthcare utilization including hospital admissions and ED visits at 12 months, and we hypothesize that utilization will be reduced in subjects who receive a pharmacy social needs intervention.

SECONDARY OUTCOMES:
Cost Analysis | 12 months
  We will calculate interventions costs combined with cost savings from reduced utilization to calculate the net costs from a health system perspective.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Black Rock Pharmacy, Buffalo, New York
  - Vital Pharmacy, Buffalo, New York
  - Riverview Professional Pharmacy, Buffalo, New York
  - Middleport Family Health Center, Middleport, New York
  - Niagara Apothecary, Niagara Falls, New York

IPD SHARING:
Plan to Share IPD: Undecided
Sharing IPD will be based on specific agreements between the institution, community partners, and the local health information exchange.

REFERENCES:
- [Background] Morse JM. Determining sample size. Qual Health Res. 2000;10(1):3-5. doi: Doi 10.1177/104973200129118183. PubMed PMID: WOS:000084385600001.
- [Background] Guest G, Bunce A, Johnson L. How many interviews are enough? An experiment with data saturation and variability. Field Method. 2006;18(1):59-82. doi: 10.1177/1525822x05279903. PubMed PMID: WOS:000242853100004.
- [Background] Daly CJ, Costello J, Mak A, Quinn B, Lindenau R, Jacobs DM. Pharmacists' perceptions on patient care services and social determinants of health within independent community pharmacies in an enhanced services network. J Am Coll Clin Pharm. 2021;4(3):288-95. doi: 10.1002/jac5.1398. PubMed PMID: WOS:000710530900005.
- [Background] LaForge K, Gold R, Cottrell E, Bunce AE, Proser M, Hollombe C, Dambrun K, Cohen DJ, Clark KD. How 6 Organizations Developed Tools and Processes for Social Determinants of Health Screening in Primary Care: An Overview. J Ambul Care Manage. 2018 Jan/Mar;41(1):2-14. doi: 10.1097/JAC.0000000000000221. PMID 28990990
- [Background] Committee on the Recommended Social and Behavioral Domains and Measures for Electronic Health Records; Board on Population Health and Public Health Practice; Institute of Medicine. Capturing Social and Behavioral Domains in Electronic Health Records: Phase 1. Washington (DC): National Academies Press (US); 2014 Jun 23. Available from http://www.ncbi.nlm.nih.gov/books/NBK195994/ PMID 24757748
- [Background] Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. Jt Comm J Qual Patient Saf. 2008 Apr;34(4):228-43. doi: 10.1016/s1553-7250(08)34030-6. PMID 18468362
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Buitron de la Vega P, Ashe EM, Xuan Z, Gast V, Saint-Phard T, Brody-Fialkin J, Okonkwo F, Power J, Wang N, Lyons C, Silverstein M, Lasser KE. A Pharmacy Liaison-Patient Navigation Intervention to Reduce Inpatient and Emergency Department Utilization Among Primary Care Patients in a Medicaid Accountable Care Organization: A Nonrandomized Controlled Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2250004. doi: 10.1001/jamanetworkopen.2022.50004. PMID 36622674
- [Background] Handley MA, Lyles CR, McCulloch C, Cattamanchi A. Selecting and Improving Quasi-Experimental Designs in Effectiveness and Implementation Research. Annu Rev Public Health. 2018 Apr 1;39:5-25. doi: 10.1146/annurev-publhealth-040617-014128. Epub 2018 Jan 12. PMID 29328873
- [Background] Daly CJ, Quinn B, Mak A, Jacobs DM. Community Pharmacists' Perceptions of Patient Care Services within an Enhanced Service Network. Pharmacy (Basel). 2020 Sep 16;8(3):172. doi: 10.3390/pharmacy8030172. PMID 32947887
- [Background] Martinez LS, Russell B, Rubin CL, Leslie LK, Brugge D. Clinical and translational research and community engagement: implications for researcher capacity building. Clin Transl Sci. 2012 Aug;5(4):329-32. doi: 10.1111/j.1752-8062.2012.00433.x. Epub 2012 Jun 28. PMID 22883610
- [Background] Wheat L, Roane TE, Connelly A, Zeigler M, Wallace J, Kim JH, Segal R. Using a pharmacist-community health worker collaboration to address medication adherence barriers. J Am Pharm Assoc (2003). 2020 Nov-Dec;60(6):1009-1014. doi: 10.1016/j.japh.2020.08.021. Epub 2020 Sep 14. PMID 32943338
- [Background] Ruiz Escobar E, Pathak S, Blanchard CM. Screening and Referral Care Delivery Services and Unmet Health-Related Social Needs: A Systematic Review. Prev Chronic Dis. 2021 Aug 12;18:E78. doi: 10.5888/pcd18.200569. PMID 34387188
- [Background] Gundersen C, Ziliak JP. Food Insecurity And Health Outcomes. Health Aff (Millwood). 2015 Nov;34(11):1830-9. doi: 10.1377/hlthaff.2015.0645. PMID 26526240
- [Background] Berkowitz SA, Hulberg AC, Hong C, Stowell BJ, Tirozzi KJ, Traore CY, Atlas SJ. Addressing basic resource needs to improve primary care quality: a community collaboration programme. BMJ Qual Saf. 2016 Mar;25(3):164-72. doi: 10.1136/bmjqs-2015-004521. Epub 2015 Nov 30. PMID 26621916
- [Background] Hood CM, Gennuso KP, Swain GR, Catlin BB. County Health Rankings: Relationships Between Determinant Factors and Health Outcomes. Am J Prev Med. 2016 Feb;50(2):129-35. doi: 10.1016/j.amepre.2015.08.024. Epub 2015 Oct 31. PMID 26526164
- [Background] Austin CP. Opportunities and challenges in translational science. Clin Transl Sci. 2021 Sep;14(5):1629-1647. doi: 10.1111/cts.13055. Epub 2021 Jul 8. PMID 33982407
- [Background] Foster AA, Daly CJ, Leong R, Stoll J, Butler M, Jacobs DM. Integrating community health workers within a pharmacy to address health-related social needs. J Am Pharm Assoc (2003). 2023 May-Jun;63(3):799-806.e3. doi: 10.1016/j.japh.2023.01.006. Epub 2023 Jan 11. PMID 36710147
- [Background] Foster AA, Daly CJ, Logan T, Logan R Jr, Jarvis H, Croce J, Jalal Z, Trygstad T, Jacobs DM. Implementation and evaluation of social determinants of health practice models within community pharmacy. J Am Pharm Assoc (2003). 2022 Jul-Aug;62(4):1407-1416. doi: 10.1016/j.japh.2022.02.005. Epub 2022 Feb 11. PMID 35256284
- [Background] Foster AA, Daly CJ, Logan T, Logan R Jr, Jarvis H, Croce J, Jalal Z, Trygstad T, Bowers D, Clark B, Moore S, Jacobs DM. Addressing social determinants of health in community pharmacy: Innovative opportunities and practice models. J Am Pharm Assoc (2003). 2021 Sep-Oct;61(5):e48-e54. doi: 10.1016/j.japh.2021.04.022. Epub 2021 May 4. PMID 34023279
- [Background] Berenbrok LA, Gabriel N, Coley KC, Hernandez I. Evaluation of Frequency of Encounters With Primary Care Physicians vs Visits to Community Pharmacies Among Medicare Beneficiaries. JAMA Netw Open. 2020 Jul 1;3(7):e209132. doi: 10.1001/jamanetworkopen.2020.9132. PMID 32667653
- [Background] Guadamuz JS, Alexander GC, Zenk SN, Qato DM. Assessment of Pharmacy Closures in the United States From 2009 Through 2015. JAMA Intern Med. 2020 Jan 1;180(1):157-160. doi: 10.1001/jamainternmed.2019.4588. PMID 31633745
- [Background] Qato DM, Zenk S, Wilder J, Harrington R, Gaskin D, Alexander GC. The availability of pharmacies in the United States: 2007-2015. PLoS One. 2017 Aug 16;12(8):e0183172. doi: 10.1371/journal.pone.0183172. eCollection 2017. PMID 28813473
- [Background] Andermann A. Screening for social determinants of health in clinical care: moving from the margins to the mainstream. Public Health Rev. 2018 Jun 22;39:19. doi: 10.1186/s40985-018-0094-7. eCollection 2018. PMID 29977645
- [Background] Fraze TK, Brewster AL, Lewis VA, Beidler LB, Murray GF, Colla CH. Prevalence of Screening for Food Insecurity, Housing Instability, Utility Needs, Transportation Needs, and Interpersonal Violence by US Physician Practices and Hospitals. JAMA Netw Open. 2019 Sep 4;2(9):e1911514. doi: 10.1001/jamanetworkopen.2019.11514. PMID 31532515
- [Background] Adler NE, Glymour MM, Fielding J. Addressing Social Determinants of Health and Health Inequalities. JAMA. 2016 Oct 25;316(16):1641-1642. doi: 10.1001/jama.2016.14058. No abstract available. PMID 27669456
- See also: The Health Leads Screening Toolkit — https://healthleadsusa.org/communications-center/resources/the-health-leads-screening-toolkit/
- See also: The Pharmacists' Patient Care Process. Joint Commission of Pharmacy Practitioners — https://jcpp.net/patient-care-process/